CLINICAL TRIAL: NCT00674648
Title: A Phase I Dose Escalation Trial of Donor T Cells Sensitized With Pentadecapeptides of the CMV-PP65 Protein for the Treatment of CMV Infections Following Allogeneic Hematopoietic Stem Cell Transplants
Brief Title: Trial of Donor T Cells Sensitized With Pentadecapeptides of the CMV-PP65 Protein for the Treatment of Cytomegalovirus (CMV) Infections Following Allogeneic Hematopoietic Stem Cell Transplants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-065
Expanded Access: NCT03010332 (No longer available)
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Cytomegalovirus Infections
Keywords: Multiple Diseases; Hematopoietic System; CMV-PP65 PROTEIN SPECIFIC T CELLS
MeSH Terms: conditions — Cytomegalovirus Infections

ARMS (1):
- 1 (Experimental): This is a non-randomized single institution phase I dose escalation trial, designed to evaluate the toxicity and anti-viral activity of CMV-pp65 peptide-specific T cell lines, generated in vitro from CMV seropositive normal HSCT and 3rd party donors, when adoptively transferred to treat recipients of these transplants who have a CMV infection or persistent CMV antigenemia and are therefore at high risk of a life-threatening CMV infection.
  Interventions: Biological: CMV-Peptide-Specific T cells

INTERVENTIONS:
Biological: CMV-Peptide-Specific T cells — In this phase I trial, five escalating dose levels will be tested. Each dose will be administered to groups of at least 3 and up to 6 patients. Dose escalation will be based on the dose limiting toxicity (DLT) observed in each treatment group (Confer Biostatistics).
  The patient groups and donors are outlined as follows: Group I will receive a single dose of 5 x 105 T cells/kg body weight/dose; Group II will receive a single dose of 1 x 106 T cells/kg/dose; and group III will receive a single dose of 2 x 106 T cells/kg/dose; group IV will receive 3 weekly doses of 1 x 106 T cells/kg/dose; group V will receive 3 weekly doses of 2 x 106 T cells/kg/dose.

SUMMARY:
The purpose of this study is to test the safety of a transfusion of specialized white cells from your transplant donor's blood, called T-cells, that have been grown and immunized against the CMV virus in the test tube. If the transplant donor is immune to CMV (ie: the donor has antibody to CMV in the blood), the T-cells will be selected and grown from the blood of the transplant donor. However, if the transplant donor is not immune to CMV, or if T-cells from the donor are not readily available, CMV-immune T-cells grown from the blood of another normal donor who is partially matched to the patients tissue type can be used. The transplant physician will explain which of these treatments is available to the patient.

This trial is called a phase I trial because phase I trials are designed to test the safety of different doses of an experimental treatment. We want to find out what effects, good and/or bad, a dose/doses of these immune T-cells will have on the patient and on the CMV infection.

Specifically, we wish to test CMV immune T-cells grown from your blood using a new method developed at our center. In this method, fragments of an important CMV protein, called CMVpp65, are chemically synthesized and then used to immunize T-cells in the test tube.

ELIGIBILITY:
Inclusion Criteria:

Prior to receiving treatment, some patients may undergo diagnostic and/or other testing of their tissue, if available, to determine if their CMV infected cells are likely to respond to treatment with CMV specific T cells. Alternatively, blood samples may be required for research tests to ascertain that the CMV-specific T-cells do not contain any cells that could react against the patient. These patients will sign a separate pre-treatment consent. If it is determined that a patient will qualify for and might benefit from infusions of CMV CTLs, he/she will go on to sign the standard treatment consent for MSKCC IRB # 05-065 and be enrolled and treated on trial, if all other eligibility criteria are met.

* Each patient must satisfy at least one of the following criteria:
* The patient must have a clinically documented condition associated with CMV (e.g. interstitial pneumonia, hepatitis, retinitis) or
* The patient must have microbiological evidence of CMV viremia or tissue invasion as attested by viral culture, or detection of CMV antigenemia or detection of levels of CMV DNA in blood or body fluids consistent with CMV infection.
* The patient's CMV infection is clinically progressing or CMV viremia is persistent or increasing (as evidenced by quantitation of CMV antigenemia or CMV DNA in the blood) despite two weeks induction therapy with antiviral drugs.
* The patient has developed CMV viremia as attested by viral culture, or detection of CMV antigenemia or detection of levels of CMV DNA in blood or body fluids while receiving prophylactic doses of antiviral drugs to prevent CMV infection post transplant. or
* the patient is unable to sustain treatment with antiviral drugs due to drug associated toxicities (e.g. myelosuppression [ANC < 1000 ul/ml without GCSF support] or nephrotoxicity [corrected creatinine clearance < than or equal to 60ml/min/1.73m2 or creatinine >2 mg/dl]).
* Because CMV infections are life-threatening and may involve the lungs, liver, gastrointestinal tract, hematopoietic and central nervous systems, and antiviral drugs may also compromise renal and hematopoietic function, dysfunctions of these organs will not affect eligibility for this protocol.

However, to be eligible, the patients should meet the following clinical criteria:

* They must have a stable blood pressure and circulation, not requiring pressor support.
* They should have adequate cardiac function as demonstrated by EKG and/or by echocardiographic evidence.
* They should have a life expectancy, even if they require respirator support, of at least 3 weeks.
* They are no age restrictions to eligibility for this protocol.

Exclusion Criteria:

* Patients requiring high doses of glucocorticosteroids (>0.5 mg/kg prednisone or its equivalent) as treatment for active (grade 2-4) acute graft vs. host disease (GVHD) or chronic GVHD.
* Patients who are moribund.
* Patients with other conditions not related to CMV infection (e.g. uncontrolled bacterial sepsis or invasive fungal infection) which are also life-threatening and which would preclude evaluation of the effects of a T cell infusion.

Donor Eligibility for Donation of Blood Lymphocytes for Generation of

Donor-Derived CMV-Specific T cells:

Adequate health for donation as determined by institutional (related donor) or NMDP (unrelated donor) guidelines. Normal donors will be evaluated for evidence of prior sensitization to CMV by CMV serology. They will also be typed for HLA A, B, C and DR. For allogeneic hematopoietic progenitor cell transplant (HSCT) recipients, the marrow transplant donor will constitute the donor of choice, since those T-cells will grow and persist in a patient who has already engrafted with a transplant from that donor. However, if the HSCT donor is CMV seronegative or not available (e.g. a cord blood transplant or an unrelated donor who has not already donated T-cells for adoptive therapy), CMV-specific T-cells generated from a seropositive donor matched for at least 2 HLA alleles shared by the patient may be used.

Normal donors fulfilling these criteria who consent to donate blood for the generation of CMV-specific T-cells for adoptive therapeutic purposes will receive a detailed clinical evaluation, including a medical history, physical examination, and serologic testing for transmissible diseases within 1 week of donation including hepBs Ag and hepatitis C antibody, HIV-1 and 2, HTLV-1 and 2, CMV (only if previously negative), VDRL, WNV, and Chagas An HIV+ donor will be rejected on medical grounds. Donors must have Hgb value > 10 gm/dl and must be capable of undergoing a single 3-6 unit leukapheresis (preferable) or a single unit of blood for T cells (for pediatric donors, no more than 5 ml/kg at any one blood draw).

A prospective donor will be informed of the purposes of this study, and its requirements. If he/she consents, the donor will be requested to provide two blood samples:

i. An initial donation of 25ml blood anticoagulated with heparin or ACD. This blood is used to establish a B cell line transformed with the B95.8 laboratory strain of EBV. This EBV+ B cell line/ (EBVBLCL) will be used as an antigen-presenting cell. When loaded with the pool of CMVpp65 pentadecapeptides, the EBVBLCL efficiently sensitize T cells from the same donors against CMV as well as EBV.

Because the establishment and testing of an EBV transformed B cell line suitable for use or as an antigen-presenting cell require 4-5 weeks of in vitro culture, it is important that this sample be obtained as early as possible for patients at risk for a CMV infection. Because patients receiving HSCT from unrelated or HLA disparate donors are particularly at risk for severe CMV infections in the first 2-3 months after transplant, this blood sample should be obtained from the donor prior to donation of the hematopoietic progenitor cell transplant whenever possible.

ii. A donation of either a single standard 2 blood volume leukapheresis collected in standard ACD anticoagulant. If it is impossible to collect a leukapheresis from some of the donors, a unit of whole blood will be acceptable. However, the AICTF (Adoptive Immune Cell Therapy Facility manufacturing the clinical grade cell products under GMP conditions in MSKCC) may only be able to generate a limited number of T cells from a unit of blood. This blood is required for isolation of the T cells to be sensitized with the pool of CMVpp65 15-mers loaded on the autologous EBVBLCL, and propagated in vitro. In addition, it is required to provide autologous feeder cells essential to sustain T-cell growth without the risk of stimulating the growth of alloreactive T-cells capable of inducing GVHD.

This donation of a leukapheresis or a unit of blood will be obtained from unrelated HSCT donors at least 2 weeks after their donation of an HSCT, or as soon as possible thereafter.

In order to limit the number of blood or leukapheresis donations that would be required of any donor, each donor will be informed of the following potential applications of the blood cells donated. The white cells contained in one leukapheresis are sufficient to grow enough T- cells to treat the three conditions below in a transplant patient:

1. The use of cells to generate CMV-specific T-cells for potential use in the treatment of the patient for whom the donor has provided an HSCT, under MSKCC IRB # 05-065.
2. The use of a fraction of the cells isolated to generate:

   1. immune T-cells specific for another virus, such as Epstein-Barr virus, that can cause lethal lymphomas in transplant recipients, and
   2. immune T-cells specific for a protein called WT-1, that is differentially expressed by malignant blood cells.

   Such T-cells could be used, under separate protocols, to treat EBV associated diseases (IRB 95-024) and/or to treat or prevent leukemia recurrence (07-055) in the patient receiving the donor's hematopoietic progenitor cell transplant.
3. The donation of the immune T-cells generated from the donor that are not used for or required by the patient for whom they were originally intended to a bank of immune cells that will be stored and maintained cryopreserved under GMP conditions in the Adoptive Immune Cell Therapy Facility at MSKCC, These stored T-cells , may be used for the treatment of other patients with CMV or EBV infections/malignancies that express HLA alleles shared by the donor.

In addition to these prospectively accrued donors, we have, since the initiation of this protocol, generated over 100 CMV-specific T-cells for patients at high risk for infection, of which far fewer patients have required treatment. Since these patients are now beyond the period of risk for CMV infection, their donors will be approached with a separate consent to allow for the use of their T cells in recipients other than the primary patients for whom they initially donated cells.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety or toxicities of escalating doses of donor-derived CMV-pp65 peptide-specific T cells. | conclusion of the study

SECONDARY OUTCOMES:
To quantitate alterations in the level of CMV antigenemia in the blood of patients with either active infection or persistent antigenemia following adoptive transfer of CMV-pp65 peptide-specific T cells. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Susan Prockop, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org